CLINICAL TRIAL: NCT06598826
Title: Graston Technique Versus Kinesio Taping on Myofascial Pain Syndrome After Neck Dissection Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hasnaa Abd-Elfatah Mohamed, Physiotherapy specialist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4648
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-07

CONDITIONS: Post Neck Dissection Surgery
Keywords: Graston technique (IASTM); Kinesiotape; Myofascial pain syndrome
MeSH Terms: conditions — Myofascial Pain Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Graston technique (Active Comparator): This group received Graston technique (IASTM) , in additional to traditional treatment (ROM exercise, strengthening exercise, and stretching exercise) 3 times per week for 1 month
  Interventions: Device: Graston technique (IASTM)
- Kinesio taping (Active Comparator): Group B includes 26 patients who received Kinesiotaping, in addition to traditional treatment (ROM exercise, strengthening exercise, and stretching exercises) 2 times per week for 1 month
  Interventions: Other: Kinesio taping

INTERVENTIONS:
Device: Graston technique (IASTM) — Group A includes 26 patients post ND who received Graston technique (IASTM) , in additional to traditional treatment (ROM exercise, strengthening exercise, and stretching exercise) for 1 month
  Other Names: Traditional treatment (ROM exercise, strengthening exercise, and stretching exercises)
  Arms: Graston technique
Other: Kinesio taping — Group B includes 26 patients who received Kinesiotaping, in addition to traditional treatment (ROM exercise, strengthening exercise, and stretching exercises) for 1 month
  Other Names: Traditional treatment (ROM exercise, strengthening exercise, and stretching exercises)
  Arms: Kinesio taping

SUMMARY:
This study was conducted to investigate the effect of Graston technique versus Kinesiotaping on myofascial pain syndrome after neck dissection surgery.

DETAILED DESCRIPTION:
Fifty two patients from both genders who had cervical Myofascial pain syndrome following a neck dissection surgery participated in this Study. Their ages ranged from 30 to 50 years. They had been selected from the National Cancer Institute, Cairo University. They were assigned randomly into two groups (A) and (B), equal in number. Group (A) received Graston technique (IASTM), in addition to traditional treatment (range of motion exercises, stretching exercises and strengthening exercises) for 12 Sessions performed in a period of 4 weeks (three times weekly). While Group (B) Received kinesiotaping, in addition to traditional treatment (range of motion exercises, stretching exercises and strengthening exercises) for 8 sessions performed in a period of 4 weeks (twice weekly). Pressure pain threshold, visual analogue scale and cervical lateral flexion and rotation were measured pre and post 4 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* The subjects were selected according to the following criteria:

The patient's ages ranged from 30 to 50 years participated in this study. Both genders participated in this study. All patients had a history of MPS at UTM from 3 to 5 months. All patients had moderate to severe pain (VAS score >4). Informed consent was obtained from every patient enrolled in the trial. All patients had myofascial pain syndrome after unilateral modified radical neck dissection surgery.

Exclusion Criteria:

* The potential participants were excluded if they meet one of the following criteria:

A wound in the affected area A cervical disk lesion Myelopathy or radiculopathy Cervical spine fracture or spondylolisthesis Rheumatoid arthritis Epilepsy or any psychological disorders Contraindications to IASTM. Contraindications to Kinesiotaping. Coagulopathy. Hemophilia or other clotting disorders.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-06-12 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Range of motion (ROM) (cervicallateralflexion) | Pretreatment, post treatment ( after 4 weeks of treatment)
  Universal Goniometer is a reliable instrument used to evaluate Range of motion in degrees
Range of motion (ROM) (cervical rotation) | Pretreatment, post treatment ( after 4 weeks of treatment)
  Universal Goniometer is a reliable instrument used to evaluate Range of motion in degrees
Pressure pain threshold | Pretreatment, post treatment ( after 4 weeks of treatment)
  Pressure Algometer with a spring is used. They maintain a peak force or pressure (KP (kilopond) = 10 N, Newton = 100 kPa (kilopascal)) until tared
Assessment of pain | Pretreatment, post treatment ( after 4 weeks of treatment)
  Vasual Analogue Scale(VAS) is used technique for assessing pain intensity , a continuous scale with a vertical or horizontal line of 100 mm, from 0 to10, whose extremes are designated "no pain" and "worst imaginable pain" (0= no pain; 10= most painful imaginable pain).

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Giza, Egypt